CLINICAL TRIAL: NCT04582604
Title: Ruxolitinib and Decitabine Intensified Conditioning Regimen for Patients With High Risk Hematological Malignancies Underwenting Allogeneic Stem Cell Transplantation
Brief Title: Ruxolitinib and Decitabine for High Risk Hematological Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2020-297-01
Record Dates: First submitted 2020-10-03; First posted 2020-10-09 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Peripheral Blood Stem Cell Transplantation
MeSH Terms: interventions — Decitabine; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib combined with Decitabine (Experimental): Ruxolitinib and Decitabine conditioning regimen All recipients in this arm received the modified Bu/Cy conditioning regimen intensified by Ruxolitinib and Decitabine. The conditioning regimen for allogeneic hematopoietic stem cell transplantation consist of ruxolitinib (35 mg bid [p.o.], days -15 to -10, diminishing to day -1), decitabine (20 mg/m2/day, days -15 to -10), cytarabine (4 g/m2/day, days -10 to -9 (for unrelated donors or haploidentical donors; and 4 g/m2/day, days -9 for sibling donors)), busulfan (0.8mg/kg, Q6h, days -8 to -6), cyclophosphamide (1.8 g/m2/day, days -5 to -4);carmustine(BCNU)(250mg/m2/day, day -3),
  Interventions: Drug: modified By/Cy conditioning regimen intensified by Ruxolitinib and Decitabine

INTERVENTIONS:
Drug: modified By/Cy conditioning regimen intensified by Ruxolitinib and Decitabine — Day -15 to -14 ： Decitabine 20 mg/m2/day, Ruxolitinib 70mg bid; Day-10： Cytarabine 1.6 g/m2/day CI (only for Haploidentical and unrelated donor), Ruxolitinib 60mg bid; Day- 9： Cytarabine 4g/m2/day CI, Ruxolitinib 60mg bid; Day- 8 to -7： Busulfan 0.8mg/kg Q6h iv, Ruxolitinib 50mg bid; Day-6: Busulfan 0.8mg/kg Q6h iv, Ruxolitinib 40mg bid; Day-5： Cyclophosphamide 1.8 g/m2/day CI, Ruxolitinib 30mg bid; Day-4： Cyclophosphamide 1.8 g/m2/day CI, Ruxolitinib 20mg bid; Day-3： Carmustine 250mg/m2/day iv, Ruxolitinib 10mg bid; Day-2： Ruxolitinib 5mg bid; Day-1： Ruxolitinib 5mg qd;
  Other Names: Ruxolitinib and Decitabine

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Ruxolitinib and Decitabine intensified Conditioning Regimen in Patients with High Risk hematological malignancies undergoing allogeneic peripheral blood stem cell transplantation.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation should be offered to eligible patients with high risk hematological malignancies whenever feasible. To further improve the outcome of transplantation patients with high risk hematological malignancies, the investigators developed a modified Bu/Cy conditioning regimen intensified by Ruxolitinib and Decitabine. In this study, the investigators tested the efficacy and feasibility of the modified Bu/Cy conditioning regimen intensified by Ruxolitinib and Decitabine in Patients with high risk hematological malignancies undergoing allogeneic peripheral blood stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/refractory acute leukemia with indications for allogeneic hematopoietic stem cell transplantation; High risk acute leukemia with indications for allogeneic hematopoietic stem cell transplantation;
2. Medium to high risk myelodysplastic syndrome, myeloproliferative disease, myelodysplastic syndrome/myeloproliferative disease, Chronic myelomonocytic leukemia;
3. Have matched sibling donors, ≥8/10 HLA matched unrelated donors or haploidentical donors
4. All patients should aged 12 to 65 years;
5. Liver function: ALT and AST≤2.5 times the upper limit of normal , bilirubin≤2 times the upper limit of normal;
6. Renal function: creatinine ≤the upper limit of normal;
7. Patients without any uncontrolled infections , without organ dysfunction or without severe mental illness;
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
9. Have signed informed consent.

Exclusion Criteria:

1. pregnant women;
2. Patients with mental illness or other states unable to comply with the protocol;
3. AML patients with t (15;17);

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants relapse as assessed by NCCN (National Comprehensive Cancer Network )criteria | 365 days after transplantation
  Defined as the proportion of participants whose underlying malignancy relapsed.

SECONDARY OUTCOMES:
DFS(disease-free survival ) | 365 days after transplantation
  DFS was defined as survival with no evidence of relapse or progression.
TRM(treatment-related mortality ) | 365 days after transplantation
  Defined as the proportion of subjects who died due to causes other than malignancy relapse.
Number of participants with aGVHD as assessed by acute graft versus host disease grading criteria (refer to Glucksberg criteria) | 100 days after transplantation
  Defined as the proportion of participants who developed acute GVHD.
Number of participants with cGVHD as assessed by chronic graft versus host disease grading criteria (refer to NIH criteria) | 365 days after transplantation
  Defined as the proportion of participants who developed chronic GVHD.
OS(overall survival ) | 365 days after transplantation
  OS was defined as the time from transplantation to death due to any cause.
GRFS (GVHD free, relapse free survival) | 365 days after transplantation
  GVHD-free, relapse-free survival (GRFS) was defined as survival with no evidence of grade III-IV acute GVHD or cGVHD requiring immunosuppressive treatment, and without disease recurrence or death from any cause during the first year after transplantation.
infection rate | 365 days after transplantation
  Defined as the proportion of participants who developed all kinds of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karjalainen R, Pemovska T, Popa M, Liu M, Javarappa KK, Majumder MM, Yadav B, Tamborero D, Tang J, Bychkov D, Kontro M, Parsons A, Suvela M, Mayoral Safont M, Porkka K, Aittokallio T, Kallioniemi O, McCormack E, Gjertsen BT, Wennerberg K, Knowles J, Heckman CA. JAK1/2 and BCL2 inhibitors synergize to counteract bone marrow stromal cell-induced protection of AML. Blood. 2017 Aug 10;130(6):789-802. doi: 10.1182/blood-2016-02-699363. Epub 2017 Jun 15. PMID 28619982
- [Background] Rampal R, Ahn J, Abdel-Wahab O, Nahas M, Wang K, Lipson D, Otto GA, Yelensky R, Hricik T, McKenney AS, Chiosis G, Chung YR, Pandey S, van den Brink MR, Armstrong SA, Dogan A, Intlekofer A, Manshouri T, Park CY, Verstovsek S, Rapaport F, Stephens PJ, Miller VA, Levine RL. Genomic and functional analysis of leukemic transformation of myeloproliferative neoplasms. Proc Natl Acad Sci U S A. 2014 Dec 16;111(50):E5401-10. doi: 10.1073/pnas.1407792111. Epub 2014 Dec 2. PMID 25516983
- [Background] Delgado-Martin C, Meyer LK, Huang BJ, Shimano KA, Zinter MS, Nguyen JV, Smith GA, Taunton J, Winter SS, Roderick JR, Kelliher MA, Horton TM, Wood BL, Teachey DT, Hermiston ML. JAK/STAT pathway inhibition overcomes IL7-induced glucocorticoid resistance in a subset of human T-cell acute lymphoblastic leukemias. Leukemia. 2017 Dec;31(12):2568-2576. doi: 10.1038/leu.2017.136. Epub 2017 May 9. PMID 28484265
- [Background] Venugopal S, Bar-Natan M, Mascarenhas JO. JAKs to STATs: A tantalizing therapeutic target in acute myeloid leukemia. Blood Rev. 2020 Mar;40:100634. doi: 10.1016/j.blre.2019.100634. Epub 2019 Oct 25. PMID 31677846
- [Background] Ding YY, Stern JW, Jubelirer TF, Wertheim GB, Lin F, Chang F, Gu Z, Mullighan CG, Li Y, Harvey RC, Chen IM, Willman CL, Hunger SP, Li MM, Tasian SK. Clinical efficacy of ruxolitinib and chemotherapy in a child with Philadelphia chromosome-like acute lymphoblastic leukemia with GOLGA5-JAK2 fusion and induction failure. Haematologica. 2018 Sep;103(9):e427-e431. doi: 10.3324/haematol.2018.192088. Epub 2018 May 17. No abstract available. PMID 29773603
- [Derived] Wei Y, Luan S, Wang L, Wang L, Li F, Jin X, Yang R, Qian K, Peng B, Tang J, Zhang H, Dou L, Liu D. Ruxolitinib and decitabine plus a busulfan-cyclophosphamide conditioning regimen for relapse prophylaxis in patients with high-risk acute myeloid leukemia or myelodysplastic syndromes. Front Immunol. 2025 Aug 18;16:1586512. doi: 10.3389/fimmu.2025.1586512. eCollection 2025. PMID 40901473
- [Derived] Wei Y, Qian K, Le N, Wang L, Li F, Luan S, Wang L, Jin X, Peng B, Wang N, Dou L, Liu D. Addition of ruxolitinib and decitabine to modified busulfan/cyclophosphamide conditioning regimen for prophylaxis relapse in high-risk acute myeloid leukemia: the phase 2 prospective study. Ann Hematol. 2024 Nov;103(11):4707-4719. doi: 10.1007/s00277-024-05972-w. Epub 2024 Sep 7. PMID 39243311